CLINICAL TRIAL: NCT03490058
Title: A Cohort for Evaluation of Open-label PrEP Delivery Among Kenyan and South African Women: The POWER Cohort
Brief Title: The Prevention Options for Women Evaluation Research (POWER) Cohort
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Desmond Tutu HIV Foundation (Other); Wits Reproductive Health and HIV Institute (Other); Kenya Medical Research Institute (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); RTI International (Other); Harvard Medical School (HMS and HSDM) (Other); University of Pittsburgh (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Connie Celum, Prof of Medicine & Global Health, Adjunct Prof of Epidemiology, SOM: Global Health, University of Washington
Other Study IDs: STUDY00000950; R01MH114544 (NIH); AID-OAA-A-15-00034 (Other Grant/Funding Number: US Agency for International Development)
Record Dates: First submitted 2018-03-19; First posted 2018-04-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: HIV/AIDS
Keywords: pre-exposure prophylaxis; young women; delivery of health care; HIV infections/prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Dried blood spots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young women: Sexually active HIV-uninfected women between 16-25 years of age will be given Truvada.
  Interventions: Drug: Truvada

INTERVENTIONS:
Drug: Truvada — A fixed dose of oral co-formulated tenofovir disoproxil fumarate (TDF)/emtricitabine (FTC) will be used as PrEP.

SUMMARY:
The POWER Cohort study is a PrEP implementation project to demonstrate Pre-exposure prophylaxis (PrEP) delivery for young women in Cape Town and Johannesburg, South Africa and Kisumu, Kenya.

DETAILED DESCRIPTION:
PrEP will be delivered to young women according to emerging national guidelines in family planning clinics (Kisumu, Kenya), youth friendly clinics (Johannesburg, South Africa), and mobile youth friendly clinics (Cape Town, South Africa). The investigators will evaluate PrEP delivery and follow cohorts of young women at each clinic location to understand PrEP uptake and use. In the Kisumu clinics, the investigators will also offer expedited partner therapy and partner HIV self-tests to women who test positive for chlamydia and/or gonorrhea. At one clinic in Johannesburg, the investigators will evaluate the use of a decision support tool to improve the decision to initiate PrEP.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-25 (16 and 17 year olds, where permissible by national regulations and local IRB approval)
* Able and willing to provide written informed consent
* Recently sexually active (defined as having had vaginal intercourse at least once in the previous three months)
* HIV uninfected based on negative HIV rapid tests, on the date of enrollment

Ages: 16 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Sexually active HIV uninfected women ages 16-25 will be recruited from family planning clinics, youth clinics, and youth outreach programs.
Sampling Method: Non-Probability Sample
Enrollment: 2255 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
Demonstrate PrEP delivery models for young women in different settings and geographies. | Up to 36 months
  Mixed methods assessment of how PrEP is implemented at the user, provider, health care facility, and community levels.

SECONDARY OUTCOMES:
PrEP initiation | Up to 36 months
  Measure the number of young women who initiate PrEP.
PrEP adherence | Up to 36 months
  Adherence by young women to PrEP. Adherence will be measured by the timing of PrEP refills and self-reported PrEP use. Blood samples for detection and quantification of PrEP levels (testing in batch) will be done for those who seroconvert to HIV and a subset who remain HIV uninfected.
HIV seroconversion | Up to 36 months
  Assess HIV incidence during PrEP use and non-use.

OTHER OUTCOMES:
Assess cost and cost-effectiveness of PrEP when delivered in public health clinics. | Up to 36 months
  Time-motion studies will be conducted to define the cost and cost effectiveness of the intervention in terms of HIV infections averted, disability-adjusted life years saved, and incremental cost-effectiveness of PrEP over routine HIV care.
Evaluate the acceptability of delivering expedited partner therapy. | Up to 36 months
  Measure the number of women who accept STI expedited partner therapy and HIV self-test kits for their partners.
Assess the effect of a decision support tool on PrEP uptake | Up to 36 months
  Using a randomized design, evaluate if a decision support tool increases PrEP uptake.
Evaluate the impact of HIV self-testing on PrEP delivery among young women receiving PrEP | Up to 12 months
  Using a pretest posttest design, evaluate the feasibility of integrating HIV self-testing into PrEP delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Connie L Celum, MD, MPH, Principal Investigator — University of Washington; Jared M Baeten, MD, PhD, Principal Investigator — University of Washington; Rachel Johnson, MPH, Study Director — University of Washington
Locations (3):
- Kenya Medical Research Institute, Kisumu, Kenya
- South Africa (2):
  - Desmond Tutu HIV Foundation, Cape Town
  - Wits Reproductive Health and HIV Institute, Johannesburg

IPD SHARING:
Plan to Share IPD: Yes
Data from the POWER Cohort Study will be available at the end of the project by contacting the Principal Investigators.

REFERENCES:
- [Derived] Katz AWK, Roberts S, Rousseau E, Khoza MN, Mogaka F, Bukusi E, Delany-Moretlwe S, Bekker LG, Morton JF, Johnson R, Baeten JM, Celum C, van der Straten A. Qualitative Analysis Using Social Maps to Explore Young Women's Experiences With Social Support of their Oral PrEP Use in Kenya and South Africa. J Assoc Nurses AIDS Care. 2023 Jan-Feb 01;34(1):45-57. doi: 10.1097/JNC.0000000000000363. Epub 2022 Sep 23. PMID 36170124
- [Derived] Celum CL, Bukusi EA, Bekker LG, Delany-Moretlwe S, Kidoguchi L, Omollo V, Rousseau E, Travill D, Morton JF, Mogaka F, O'Malley G, Barnabee G, van der Straten A, Donnell D, Parikh UM, Kudrick L, Anderson PL, Haberer JE, Wu L, Heffron R, Johnson R, Morrison S, Baeten JM; POWER Study Team. PrEP use and HIV seroconversion rates in adolescent girls and young women from Kenya and South Africa: the POWER demonstration project. J Int AIDS Soc. 2022 Jul;25(7):e25962. doi: 10.1002/jia2.25962. PMID 35822945
- [Derived] Roche SD, Barnabee G, Omollo V, Mogaka F, Odoyo J, Bukusi EA, Morton JF, Johnson R, Celum C, Baeten JM, O'Malley G. Implementation strategies for integrating pre-exposure prophylaxis for HIV prevention and family planning services for adolescent girls and young women in Kenya: a qualitative study. BMC Health Serv Res. 2022 Mar 30;22(1):422. doi: 10.1186/s12913-022-07742-8. PMID 35354456
- [Derived] Omollo V, Bukusi EA, Kidoguchi L, Mogaka F, Odoyo JB, Celum C, Morton J, Johnson R, Baeten JM. A Pilot Evaluation of Expedited Partner Treatment and Partner Human Immunodeficiency Virus Self-Testing Among Adolescent Girls and Young Women Diagnosed With Chlamydia trachomatis and Neisseria gonorrhoeae in Kisumu, Kenya. Sex Transm Dis. 2021 Oct 1;48(10):766-772. doi: 10.1097/OLQ.0000000000001430. PMID 33859147